CLINICAL TRIAL: NCT00204412
Title: Effectiveness of Flax Lignan and Exercise Training for Improving Lipid Profiles
Brief Title: Exercise and Flax-Based Nutritional Supplementation for Lowering Cholesterol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 686868
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Metabolic Syndrome; Osteoporosis
Keywords: Cholesterol; High density lipoprotein; Low density lipoprotein; Triglyceride; Glucose; Exercise; Fitness; Flax; Lignan; Phytoestrogen; bone
MeSH Terms: conditions — Metabolic Syndrome; Osteoporosis; Motor Activity | interventions — Exercise; Walking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): flax lignan
  Interventions: Dietary Supplement: Flax lignan; Behavioral: Exercise (walking)
- 2 (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Flax lignan

INTERVENTIONS:
Dietary Supplement: Flax lignan — 543 mg SDG per day
  Other Names: Archer Daniels Midland
Behavioral: Exercise (walking) — walking 45 minutes per day 5 days per week
  Arms: 1

SUMMARY:
The purpose of our study is to use a flaxseed-based nutritional supplement in combination with exercise training (walking) for improving cholesterol levels. We hypothesize that exercise training will improve cholesterol profile and that adding supplementation with a flaxseed nutritional supplement will further improve cholesterol profile.

DETAILED DESCRIPTION:
Flax supplementation and exercise training each have small beneficial effects for improving blood lipid profile and reducing cardiovascular disease risk. Flax lignan, a phytoestrogen found in flaxseed is thought to be the active compound responsible for the cholesterol-lowering effect of flaxseed. Our purpose is to combine an exercise training program (walking) with flax lignan supplementation for improving blood lipid profile.

Comparisons: Walking (6 days per week) plus flax lignan (500 mg per day) compared to walking plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older

Exclusion Criteria:

* Currently taking medication for cholesterol
* Smoker
* Diabetic
* Gastrointestinal disease
* Females on hormone replacement therapy
* Currently taking a flaxseed supplement
* Currently engaged in vigorous exercise training

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-03; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
metabolic syndrome score | 6 months

SECONDARY OUTCOMES:
Total cholesterol at 2, 4, and 6 months | 6 months
High density lipoprotein at 2, 4, and 6 months | 6 months
Low density lipoprotein at 2, 4, and 6 months | 6 months
Triglycerides at 2, 4, and 6 months | 6 months
Blood glucose at 2, 4, and 6 months | 6 months
Body composition at 6 months | 6 months
Aerobic fitness at 6 months | 6 months
Waist Girth at 6 months | 6 months
Body mass index at 6 months | 6 months
Lumbar spine bone mineral density at 6 months | 6 months
Proximal femur bone mineral density at 6 months | 6 months
Whole body bone mineral density at 6 months | 6 months
Trunk fat skinfolds at 6 months | 6 months
inflammatory cytokines | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Chilibeck, PhD, Principal Investigator — University of Saskatchewan; H J Biem, MD, Study Director — University of Saskatchewan; Lisa Paus-Jenssen, MD, Study Director — University of Saskatchewan; Susan Whiting, PhD, Study Director — University of Saskatchewan; Punam Pahwa, PhD, Study Director — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada